CLINICAL TRIAL: NCT01027650
Title: Safety and Efficacy of AGN208397 in the Treatment of Macular Edema Associated With Retinal Vein Occlusion (RVO)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 208397-001
Record Dates: First submitted 2009-12-04; First posted 2009-12-08 (Estimated); Results first posted 2014-04-29 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-03

CONDITIONS: Macular Edema; Retinal Vein Occlusion
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Stage 1 Cohort 1 (Experimental): AGN208397 intravitreal injection 75 ug on Day 1.
  Interventions: Drug: AGN208397 intravitreal injection
- Stage 1 Cohort 2 (Experimental): AGN208397 intravitreal injection 300 ug on Day 1.
  Interventions: Drug: AGN208397 intravitreal injection
- Stage 1 Cohort 3 (Experimental): AGN208397 intravitreal injection 600 ug on Day 1.
  Interventions: Drug: AGN208397 intravitreal injection
- Stage 1 Cohort 4 (Experimental): AGN208397 intravitreal injection 900 ug on Day 1.
  Interventions: Drug: AGN208397 intravitreal injection
- Stage 2 Arm 1 (Experimental): AGN208397 intravitreal injection 600 ug on Day 1.
  Interventions: Drug: AGN208397 intravitreal injection
- Stage 2 Arm 2 (Experimental): AGN208397 intravitreal injection 450 ug on Day 1.
  Interventions: Drug: AGN208397 intravitreal injection
- Stage 2 Arm 3 (Experimental): AGN208397 intravitreal injection 300 ug on Day 1.
  Interventions: Drug: AGN208397 intravitreal injection
- Stage 2 Arm 4 (Active Comparator): Dexamethasone 700 ug intravitreal implant on Day 1.
  Interventions: Drug: dexamethasone intravitreal implant

INTERVENTIONS:
Drug: AGN208397 intravitreal injection — AGN208397 intravitreal injection on Day 1.
  Arms: Stage 1 Cohort 1; Stage 1 Cohort 2; Stage 1 Cohort 3; Stage 1 Cohort 4; Stage 2 Arm 1; Stage 2 Arm 2; Stage 2 Arm 3
Drug: dexamethasone intravitreal implant — Dexamethasone 700 ug intravitreal implant on Day 1.
  Other Names: Ozurdex®
  Arms: Stage 2 Arm 4

SUMMARY:
This study will evaluate the safety and efficacy of a single intravitreal injection of AGN208397 to treat Macular Edema associated with Retinal Vein Occlusion. This study is being conducted in two stages: Stage 1 will enroll approximately 21 subjects who will receive a single open label intravitreal injection of either 75 ug, 300 ug, 600 ug or 900 ug of AGN208397 and be followed for 12 months post treatment; based on Stage 1 results, Stage 2 will enroll approximately 96 subjects who will receive a single masked intravitreal injection of one of three doses of AGN208397 or Ozurdex® and be followed for 12 months post treatment.

ELIGIBILITY:
Inclusion Criteria:

* macular edema due to retinal vein occlusion
* visual acuity in the study eye between 20/320 to 20/40

Exclusion Criteria:

* cataract surgery or Lasik within 3 months prior to study Day 1 or anticipated need for cataract surgery during study period (12 months)
* use of injectable drugs in the study eye within 2 months prior to day 1
* active eye infection in either eye
* visual acuity in the non-study eye of 20/200 or worse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2010-03; Primary Completion 2012-04 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (5):
- Phoenix, Arizona, United States
- East Melbourne, Victoria, Australia
- London, Ontario, Canada
- Tel Aviv, Israel
- Cape Town, South Africa

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Doses for Stage 2 were selected based on the safety and pharmacodynamic results from Stage 1. No patients in Stage 1 were enrolled in Stage 2.
Period: Overall Study
Arm/Group | Stage 1 Cohort 4 | Stage 1 Cohort 3 | Stage 1 Cohort 2 | Stage 1 Cohort 1 | Stage 2 Arm 1 | Stage 2 Arm 2 | Stage 2 Arm 3 | Stage 2 Arm 4
Started | 6 | 6 | 6 | 3 | 25 | 26 | 25 | 24
Completed | 6 | 6 | 6 | 3 | 23 | 24 | 24 | 24
Not Completed | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0
Not completed — Personal Reasons | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stage 1 Cohort 4 | Stage 1 Cohort 3 | Stage 1 Cohort 2 | Stage 1 Cohort 1 | Stage 2 Arm 1 | Stage 2 Arm 2 | Stage 2 Arm 3 | Stage 2 Arm 4 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 3 | 25 | 26 | 25 | 24 | 121
Age, Customized [Number; unit: Participants]
  <45 years | 1 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 10
  Between 45 and 65 years | 3 | 4 | 4 | 0 | 8 | 10 | 11 | 9 | 49
  >65 years | 2 | 2 | 2 | 3 | 17 | 13 | 11 | 12 | 62
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 1 | 10 | 11 | 13 | 12 | 54
  Male | 4 | 4 | 3 | 2 | 15 | 15 | 12 | 12 | 67

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Month 1 in Retinal Thickness in the Study Eye During Stage 1
Description: Retinal thickness is assessed by optical coherence tomography (OCT) in the study eye. The retina is the light-sensitive part of the eye. OCT is a laser-based, noninvasive, diagnostic system providing high-resolution, three-dimensional images of the retina. A negative change from baseline indicates an improvement.
Time Frame: Baseline, Month 1
Population: Safety Population: all patients who received study treatment
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | Stage 1 Cohort 4 | Stage 1 Cohort 3 | Stage 1 Cohort 2 | Stage 1 Cohort 1
Number analyzed (Participants) | 6 | 6 | 6 | 3
Microns
  Baseline | 500.2 (197.58) | 495.8 (163.13) | 499.5 (158.33) | 468.3 (24.34)
  Change from Baseline at Month 1 | -234.3 (200.23) | -210.5 (173.69) | -256.2 (102.61) | -206.7 (96.40)

2. Primary Outcome: Change From Baseline at Month 1 in Retinal Thickness in the Study Eye During Stage 2
Description: Retinal thickness is assessed by OCT in the study eye. The retina is the light-sensitive part of the eye. OCT is a laser-based, noninvasive, diagnostic system providing high-resolution, three-dimensional images of the retina. A negative change from baseline indicates an improvement.
Time Frame: Baseline, Month 1
Population: Per Protocol Population: all randomized and treated qualified patients with baseline and at least one post-baseline data for retinal thickness or BCVA in the study eye
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | Stage 2 Arm 1 | Stage 2 Arm 2 | Stage 2 Arm 3 | Stage 2 Arm 4
Number analyzed (Participants) | 23 | 25 | 21 | 23
Microns
  Baseline | 612.6 (166.15) | 637.8 (203.69) | 597.9 (217.54) | 679.7 (237.20)
  Change from Baseline at Month 1 | -298.5 (174.59) | -314.1 (169.35) | -307.0 (217.98) | -317.3 (212.51)

3. Primary Outcome: Change From Baseline at Month 1 in Best Corrected Visual Acuity (BCVA) in the Study Eye During Stage 1
Description: BCVA is measured using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved.
Time Frame: Baseline, Month 1
Population: Safety Population: all patients who received study treatment
Measure: Mean (Standard Deviation); unit: Number of Letters Read Correctly
Arm/Group | Stage 1 Cohort 4 | Stage 1 Cohort 3 | Stage 1 Cohort 2 | Stage 1 Cohort 1
Number analyzed (Participants) | 6 | 6 | 6 | 3
Number of Letters Read Correctly
  Baseline | 54.5 (16.13) | 50.2 (14.12) | 59.7 (6.62) | 53.0 (9.54)
  Change from Baseline at Month 1 | 10.0 (8.72) | 11.7 (7.17) | 8.7 (4.84) | 9.7 (2.31)

4. Primary Outcome: Change From Baseline at Month 1 in BCVA in the Study Eye During Stage 2
Description: as for outcome 3
Time Frame: Baseline, Month 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Number of Letters Read Correctly
Arm/Group | Stage 2 Arm 1 | Stage 2 Arm 2 | Stage 2 Arm 3 | Stage 2 Arm 4
Number analyzed (Participants) | 23 | 25 | 22 | 23
Number of Letters Read Correctly
  Baseline | 49.5 (12.88) | 47.6 (13.60) | 58.2 (12.89) | 50.5 (14.27)
  Change from Baseline at Month 1 | 12.0 (9.38) | 12.5 (12.74) | 14.0 (12.35) | 11.0 (11.99)

5. Secondary Outcome: Change From Baseline at Month 12 in Retinal Thickness in the Study Eye During Stage 1
Description: as for outcome 2
Time Frame: Baseline, Month 12
Population: Safety Population: all patients who received study treatment
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | Stage 1 Cohort 4 | Stage 1 Cohort 3 | Stage 1 Cohort 2 | Stage 1 Cohort 1
Number analyzed (Participants) | 6 | 6 | 6 | 3
Microns
  Baseline | 500.2 (197.58) | 495.8 (163.13) | 499.5 (158.33) | 468.3 (24.34)
  Change from Baseline at Month 12 (N=3, 3, 3, 3) | -221.7 (208.33) | -173.0 (145.01) | -239.7 (121.33) | -167.7 (96.72)

6. Secondary Outcome: Change From Baseline at Month 12 in Retinal Thickness in the Study Eye During Stage 2
Description: as for outcome 2
Time Frame: Baseline, Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | Stage 2 Arm 1 | Stage 2 Arm 2 | Stage 2 Arm 3 | Stage 2 Arm 4
Number analyzed (Participants) | 23 | 25 | 21 | 23
Microns
  Baseline | 612.6 (166.15) | 637.8 (203.69) | 597.9 (217.54) | 679.7 (237.20)
  Change from Baseline at Month 12 | -252.8 (177.09) | -218.0 (166.57) | -208.2 (200.48) | -169.1 (213.50)

7. Secondary Outcome: Change From Baseline at Month 12 in BCVA in the Study Eye During Stage 1
Description: as for outcome 3
Time Frame: Baseline, Month 12
Population: Safety Population: all patients who received study treatment
Measure: Mean (Standard Deviation); unit: Number of Letters Read Correctly
Arm/Group | Stage 1 Cohort 4 | Stage 1 Cohort 3 | Stage 1 Cohort 2 | Stage 1 Cohort 1
Number analyzed (Participants) | 6 | 6 | 6 | 3
Number of Letters Read Correctly
  Baseline | 54.5 (16.13) | 50.2 (14.12) | 59.7 (6.62) | 53.0 (9.54)
  Change from Baseline at Month 12 (N=6, 5, 6, 3) | 14.2 (15.30) | 0.8 (24.88) | 11.0 (7.43) | 14.0 (5.29)

8. Secondary Outcome: Change From Baseline at Month 12 in BCVA in the Study Eye During Stage 2
Description: as for outcome 3
Time Frame: Baseline, Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Number of Letters Read Correctly
Arm/Group | Stage 2 Arm 1 | Stage 2 Arm 2 | Stage 2 Arm 3 | Stage 2 Arm 4
Number analyzed (Participants) | 23 | 25 | 22 | 23
Number of Letters Read Correctly
  Baseline | 49.5 (12.88) | 47.6 (13.60) | 58.2 (12.89) | 50.5 (14.27)
  Change from Baseline at Month 12 | 8.0 (13.55) | 10.2 (17.22) | 12.4 (14.31) | 5.0 (11.18)

ADVERSE EVENTS:
Description: Adverse events (AEs) and serious adverse events (SAEs) are reported by treatment group assigned during Stage 1 and Stage 2. The Safety Population consisted of all patients who received the study treatment, and was used to assess AEs and SAEs.
Arm/Group | Stage 1 Cohort 4 | Stage 1 Cohort 3 | Stage 1 Cohort 2 | Stage 1 Cohort 1 | Stage 2 Arm 1 | Stage 2 Arm 2 | Stage 2 Arm 3 | Stage 2 Arm 4
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6 | 1/6 | 0/3 | 4/25 | 4/26 | 2/25 | 3/24
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 3/3 | 25/25 | 26/26 | 25/25 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Stage 1 Cohort 4 (N=6) | Stage 1 Cohort 3 (N=6) | Stage 1 Cohort 2 (N=6) | Stage 1 Cohort 1 (N=3) | Stage 2 Arm 1 (N=25) | Stage 2 Arm 2 (N=26) | Stage 2 Arm 3 (N=25) | Stage 2 Arm 4 (N=24)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastric Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0/4 | 0/4 | 0/3 | 0/2 | 0/15 | 1/15 | 0/12 | 0/12
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Facet Joint Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pseudoendophthalmitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrioventricular Block Second Degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial Ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Stage 1 Cohort 4 (N=6) | Stage 1 Cohort 3 (N=6) | Stage 1 Cohort 2 (N=6) | Stage 1 Cohort 1 (N=3) | Stage 2 Arm 1 (N=25) | Stage 2 Arm 2 (N=26) | Stage 2 Arm 3 (N=25) | Stage 2 Arm 4 (N=24)
Intraocular Pressure Increased (Investigations) | 4 | 3 | 1 | 0 | 6 | 8 | 9 | 5
Conjunctival Haemorrhage (Eye disorders) | 2 | 3 | 2 | 1 | 6 | 6 | 4 | 9
Cataract (Eye disorders) | 2 | 2 | 1 | 0 | 1 | 4 | 1 | 1
Retinal Haemorrhage (Eye disorders) | 2 | 1 | 4 | 2 | 4 | 7 | 6 | 3
Blood Urea Increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood Glucose Increased (Investigations) | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 1
Protein Urine Present (Investigations) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Eye Pain (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 3
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 4
Macular Fibrosis (Eye disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Ocular Hypertension (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 3 | 1 | 1
Cystoid Macular Oedema (Eye disorders) | 1 | 0 | 3 | 0 | 1 | 1 | 3 | 3
Eye Pruritus (Eye disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Medication Residue (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Vitreous Floaters (Eye disorders) | 1 | 0 | 0 | 1 | 4 | 7 | 3 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arteriosclerotic Retinopathy (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blepharitis (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye Swelling (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mean Cell Haemoglobin Concentration Decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection Bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal Pruritus (Reproductive system and breast disorders) | 1/2 | 0/2 | 0/3 | 0/1 | 0/10 | 0/11 | 0/13 | 0/12
Visual Acuity Reduced (Eye disorders) | 0 | 3 | 1 | 0 | 3 | 5 | 0 | 3
Vitreous Detachment (Eye disorders) | 0 | 2 | 1 | 1 | 2 | 0 | 1 | 5
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Cataract subcapsular (Eye disorders) | 0 | 1 | 1 | 0 | 1 | 2 | 3 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 2 | 2 | 1 | 0
Foreign Body Sensation in Eyes (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Macular Oedema (Eye disorders) | 0 | 1 | 1 | 0 | 3 | 5 | 5 | 11
Photophobia (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
White Blood Cells Urine Positive (Investigations) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 2
Alanine Aminotransferase Increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 1 | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood Bilirubin Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood Pressure Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival Hyperaemia (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Conjunctival Oedema (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Facial Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 3 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Iris Adhesions (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Iris Neovascularisation (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 3 | 2 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Optic Nerve Infarction (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Posterior Capsule Opacification (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Retinal Aneurysm (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Retinal Neovascularisation (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Seasonal Allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous Opacities (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 0 | 2 | 1 | 3 | 0 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood Triglycerides Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diabetic Retinopathy (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry Eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1
Macular Cyst (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Macular Degeneration (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Nitrite Urine Present (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Retinal Exudates (Eye disorders) | 0 | 0 | 1 | 0 | 4 | 3 | 4 | 3
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urine Leukocyte Esterase Positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0/4 | 0/4 | 0/3 | 1/2 | 0/15 | 1/15 | 0/12 | 1/12
Blepharal Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cataract Nuclear (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Localised Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0
Pterygium (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Retinal pigment epitheliopathy (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Retinal Vein Occlusion (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0
Angina Pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Blood Cholesterol Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Optic Disc Haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Vulvovaginal Mycotic Infection (Infections and infestations) | 0/2 | 0/2 | 0/3 | 0/1 | 0/10 | 0/11 | 1/13 | 0/12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Anterior Chamber Cell (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anterior Chamber Angle Neovascularisation (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anterior Chamber Flare (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Anterior Chamber Inflammation (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Lenticular Opacities (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.